CLINICAL TRIAL: NCT05486221
Title: Atrial Imaging and Cardiac Rhythm In Embolic Stroke. Atrial Fibrilation, Parafibrillatory Electrocardiographic Patterns and Advanced Echocardiography for Left Atrial Evaluation in Cryptogenic Stroke.
Brief Title: Atrial Imaging and Cardiac Rhythm In Embolic Stroke
Acronym: ARIES
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Collaborators: Hospital Universitario La Paz (Other); Proyecto Ictus- Grupo Estudio Enfermedades CerebroVasculares de la Sociedad Española de Neurología (Unknown)
Responsible Party: Sponsor
Other Study IDs: PI-4509
Record Dates: First submitted 2022-08-02; First posted 2022-08-03 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-05

CONDITIONS: Cryptogenic Stroke; Atrial Fibrillation; Atrial Dilatation; Stroke, Ischemic
MeSH Terms: conditions — Ischemic Stroke; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cryptogenic stroke patients: Patients with an acute ischemic stroke of cryptogenic origin with a previous negative work-up that includes: blood analysis, brain CT / MRI, angio-TC / angio-MRI, brain vessel ultrasound, ECG, 24h ECG-holter, echocardiography).
  Interventions: Other: Extensive cardiologic work-up

INTERVENTIONS:
Other: Extensive cardiologic work-up — Specific 3D and 2D echocardiography measuring left ventricule and left atrial dimensions as well as longitudinal strain. 30 day prolonged ECG monitoring.

SUMMARY:
The ARIES study is an observational study in which patients with a recent acute ischemic stroke of cryptogenic aetiology are consecutively enrolled in order to perform a extensive cardiologic work-up. The main objective is to study parameters that could predict arrythmias on prolonged monitoring and also echocardiographic parameters of left atrial disfunction that could predict the presence of a hidden atrial fibrilation and recurrent ischemic events in patients with cryptogenic stroke.

DETAILED DESCRIPTION:
Cerebrovascular diseases are the second most frequent cause of death in the general population, representing a 10% of global death. In order to prevent recurrent strokes, it is crucial to identify the underlying cause to administrate the best treatment in secondary prevention. Cryptogenic strokes are those in which the etiology remains unknown despite performing an extensive work-up; they represent between 20-62% of strokes. Occult atrial fibrilation is thought underlie up to 40% of cryptogenic strokes; it has also reciently been postulated that other left atrial arrythmias (parafibrilatory status) and left atrial markers of disfunction could represent a cardiac source of emboli.

Tha hypothesis of the ARIES study is that an extensive cardiologic work-up (advanced echocardiography measuring strain /stain rate and 3D echo and a 30 day continuos ECG monitoring) would detect atrial disfunction, parafibrilatory status and atrial fibrilation in patients with cryptogenic stroke, and that patients with these findings could have more stroke recurrences. This study is designed as a prospective observational unicentric study that includes patients with cryptogenic stroke in a consecutive matter in La Paz University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients addmitted to the Neurology service at La Paz University Hospital with a recent diagnosis of cryptogenic stroke considered non-lacunar and where no other reasonable diagnosis is suspected.
* Signed informed consent.

Exclusion Criteria:

* Presence of large vessel atheromatosis with >50% estenosis, or <50% but with two or more vascular risk factors (age > 50 years old, hipertension, diabetes mellitus, dyslipidemia, smoker).
* Patients with a un favorable clinical situation or dependance who will not benefit from the study or those that could not fullfill study visits and procedures.
* Patients in which an embolic arrythmia has already been demonstrated

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 50 years old addmitted to the neurology ward in La Paz University Hospital with a recent diagnosis of cryptogenic ischemic stroke.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-12-17 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Analyze frequency of parafibrilatory status in cryptogenic stroke patients | 30 days
  Analyze the frequency of parafibrilatory status defined as > 3000 atrial ectopic beats per day or more or >2 "micro-AF" episodes per day (fibrillatory burst <30 seconds without a monomorphic P wave ) on 30 day ECG monitoring
Analyze frequency of ecocardiographic parameters of atrial disfunction | During hospitalization
  Dimensions and function of left atrium, telesystolic volume, left auricular ejection fraction, atrial longitudinal strain in 3 phases (reservoir, conduict, contractile)
Frequency of detection of atrial fibrilation | 60 days
  Frequency of detection of atrial fibrilation lasting for more than 30 seconds on two 30 day ECG monitoring.
Correlation of parafibrilatory state and echocardiographic parameters of atrial disfunction with the probability of detection of atrial fibrilation. | 30 days
  Correlation of parafibrilatory state and echocardiographic parameters of atrial disfunction with the probability of detection of atrial fibrilation of more than 30 seconds of duration in 30-day ECG monitoring.
Correlation of parafibrilatory state and echocardiographic parameters of atrial disfunction with the probability of stroke recurrence. | At 3 months and 1 year.
  Correlation of parafibrilatory state and echocardiographic parameters of atrial disfunction with the probability of stroke recurrence in patients without documented atrial fibrilation.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Rigual Bobillo, MD, Principal Investigator — Hospital Universitario La Paz
Locations (1):
- La Paz University Hospital, Madrid, Spain